CLINICAL TRIAL: NCT00737035
Title: Testing an IHCA for Guardians of Survivors of Intraparental Homicide
Brief Title: Effectiveness of a Web-based Intervention for Guardians of Children Whose One Parent Has Murdered the Other
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Kathryn Laughon, PhD RN, University of Virginia School of Nursing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2008-0130-00; R21MH082197 (NIH); 1R21MH082197-01A1 (NIH); DDTR B3-PDS
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Intimate Partner Homicide; Parental Homicide; Guardians of Child Survivors of Parental Homicide; Post-Traumatic Stress Disorder; Uxoricide Project
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1-Intervention (Experimental): For 16 weeks, participants will have access to an interactive healthcare communication application (IHCA).
  Interventions: Behavioral: Interactive Healthcare Communication Application
- 2- Control (Active Comparator): For 16 weeks, participants will have access to generally available Internet-based information about parenting, trauma, and child development.
  Interventions: Behavioral: Control Web sites

INTERVENTIONS:
Behavioral: Interactive Healthcare Communication Application — The IHCA is an Internet-based tool that integrates multiple resources for guardians of survivors of interparental homicide. The IHCA will have six components: (1) an instant library of articles on topics of interest; (2) a resource directory of both national and local support and service organizations; (3) access to a peer communication system; (4) a Frequently Asked Questions section, updated with responses to user generated questions; (5) an "Ask an Expert" system staffed by researchers; and (6) personal stories of others dealing with IPH.
  Other Names: IHCA
  Arms: 1-Intervention
Behavioral: Control Web sites — Only publicly available Web sites on parenting, child development, and trauma will be used.
  Arms: 2- Control

SUMMARY:
This study will determine whether a specialized Web site geared for the guardians of children whose one parent has murdered the other can increase guardian capabilities, reduce guardian stress, and improve child behavior and mental health.

DETAILED DESCRIPTION:
Intraparental homicide (IPH), when one parent kills the other, leaves approximately 4,000 children bereaved each year, adding to a total of 70,000 currently in the United States. Although few studies have focused on this phenomenon, available data indicate children of IPH suffer short- and long-term mental health consequences, including post-traumatic stress disorder (PTSD). Prior research also indicates that guardians, often family members under stress themselves, do not know how to help the children. No interventions directed at guardians of child survivors of IPH are found in scientific and clinical literature. Use of a specialized Web site called an Interactive Healthcare Communication Application (IHCA) has been found effective in treating multiple health conditions, including breast cancer in women and asthma in children. This study aims to refine an IHCA Web site for use by guardians of child survivors of IPH, to determine the safety and effectiveness of this Web site, and to determine how it is used by targeted guardians.

In the first phase of this study researchers will develop the IHCA based on feedback from a small focus group of guardians of child survivors of IPH. Then guardians of survivors of IPH up to 16 years old will be randomly assigned either to receive access to the IHCA created for them or to have access only to generally available Internet information. The IHCA will have six components: (1) an Instant Library of articles on topics of interest; (2) a resource directory of both national and local support and service organizations; (3) access to a peer communication system; (4) a Frequently Asked Questions section, updated with responses to user generated questions; (5) an "Ask an Expert" system staffed by researchers; and (6) personal stories of others dealing with IPH. Participants with access to the IHCA will receive print and phone instructions explaining the Web site and have their usage monitored by tracking software. Those in the control group will be directed to a Web site linking to publically available, pre-existing support Web sites. After 16 weeks of unlimited access to the IHCA or control group Web sites from their home computers, all participants will complete four evaluation reviews: the Family Crisis Oriented Personal Evaluation Scales, the Parenting Stress Index, the Child Behavior Checklist, and the Child PTSD Inventory - Parent.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and read English at a 7th grade level
* Guardian of a child survivor of parental homicide aged 0 to 16 years

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Family Crisis Oriented Personal Evaluation Scales (F-COPES) | Measured at 16 weeks

SECONDARY OUTCOMES:
Parenting Stress Index (PSI) | Measured at 16 weeks
Child Behavior Checklist (CBCL/6-18) Parent form | Measured at 16 weeks
Child PTSD Inventory-Parent (CPTSDI-P): | Measured at 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn S. Laughon, PhD RN, Principal Investigator — University of Virginia School of Nursing
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Laughon K, Steeves RH, Parker B, Knopp A, Sawin EM. Forgiveness, and other themes, in women whose fathers killed their mothers. ANS Adv Nurs Sci. 2008 Apr-Jun;31(2):153-63. doi: 10.1097/01.ANS.0000319565.68760.4d. PMID 18497591
- [Background] Steeves R, Laughon K, Parker B, Weierbach F. Talking about talk: the experiences of boys who survived intraparental homicide. Issues Ment Health Nurs. 2007 Aug;28(8):899-912. doi: 10.1080/01612840701493576. PMID 17729173